CLINICAL TRIAL: NCT00977951
Title: A Single Centre, Double-blind, Methodology Trial to Investigate the Genomic Changes Associated With Accelerated Healing and Reduced Scarring of Small Wounds Using RN1001 in Healthy Male Subjects
Brief Title: Genomic Changes Associated With the Use of Intradermal Avotermin (Juvista) in Small Wounds in Healthy Male Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RN1001-319-1004
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing
Keywords: Cicatrix; Scar; Avotermin; Juvista; RN1001; TGF beta 3
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Transforming Growth Factor beta3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal avotermin (Experimental)
  Interventions: Drug: Intradermal avotermin
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle); Drug: Placebo

INTERVENTIONS:
Drug: Intradermal avotermin — 50 ng/100 ul avotermin administered intradermally prior to wounding (day 0) and again 24 h later on day 1. Wounds were dosed again prior to wound excision on day 3 and again on day 4
  Other Names: Juvista; RN1001; TGF beta 3
  Arms: Intradermal avotermin
Drug: Intradermal avotermin — 50 ng/100 ul avotermin administered intradermally prior to wounding (day 0) and again 24 h later on day 1. Wounds were dosed again prior to wound excision on day 5 and again on day 6
  Other Names: Juvista; RN1001; TGF beta 3
  Arms: Intradermal avotermin
Drug: Placebo (vehicle) — Placebo administered intradermally prior to wounding (day 0) and again 24 h later on day 1. Wounds were dosed again prior to wound excision on day 3 and again on day 4
  Arms: Placebo (vehicle)
Drug: Placebo — 50 ng/100 ul avotermin administered intradermally prior to wounding (day 0) and again 24 h later on day 1. Wounds were dosed again prior to wound excision on day 5 and again on day 6
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to further determine the safety and toleration of intradermal avotermin (Juvista), confirm accelerated healing and investigate genomic expression profiles

DETAILED DESCRIPTION:
Subjects were allocated to two groups. Group 1 had scheduled visits on Day 0, 1, 3 and 4 while group 2 were scheduled for Day 0, 1, 5 and 6. Follow-up post-trial safety assessments were made on Day 10-20.

On Day 0 each subject received a total of four 1cm incision wounds; two each to the upper, inner aspect of each arm. Two areas for incision were marked out on the inner aspect of each upper arm and anaesthetised before intradermal injection of Juvista or placebo. One incision site on each arm received a dose of 50ng/100μl Juvista and the other incision site received Placebo. Following injection a full thickness 1cm incision was made along the marked site.

On Day 1 all subjects were re-injected with the same dose of Juvista or placebo, 100μl to each wound margin (200μl per wound site).

On Day 3 subjects in Group 1 were re-dosed with 200μl Juvista or Placebo per site (100μl per linear cm approximated wound margin) in Arm 1. These sites were then excised with an elliptical excision. On Day 4 the same subjects received another dose of Juvista or placebo as before.

Subjects in group 2 received the same treatment to their Arm 1 as those in group 1, except on Day 5 and 6.

All wounds were monitored and photographed at two monthly intervals over the course of 6 months. At month 6, all incision sites on Arm 2 for both groups were excised.

All excised wounds were snap frozen for genomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Caucasian, male subjects aged 18-45 years inclusive.
* Weight between 60-100 kg and a BMI within the permitted range for their height using Quetelet's index - weight (kg)/height²(m). The permitted index is between 18-28.
* Non-smokers, or ex-smokers that have not smoked for at least 3 months prior to screening.

Exclusion Criteria:

* Subjects who have history or evidence of hypertrophic or keloid scarring or with tattoos or previous scars in the area to be biopsied.
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring.
* Subjects who have evidence of any past or present clinically significant disease, particularly coagulation disorders, immuno-mediated conditions and skin diseases and allergies, such as clinically significant eczema.
* Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine or allergy to surgical dressings to be used in this trial.
* Subjects with any clinically significant abnormality following review of pre-trial laboratory data and physical examination.
* Subjects who are taking, or have taken, certain prescribed or investigational drugs in the three weeks prior to Day 0 and in particular topical or systemic steroids, anti-inflammatory and anti-coagulant drugs. Certain drugs are not excluded in this trial. These include OTC analgesics including paracetamol and codeine, vitamin and mineral supplements and OTC cold remedies.
* Subjects who drink more than 28 units of alcohol per week (1 unit = 1/2 pint of beer (285mls) or 25ml of spirits or 1 glass of wine).
* Subjects who have evidence of drug abuse.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen or hepatitis C antibody. Subjects with previous vaccination against Hepatitis B are not excluded per se.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B core antibody and who show less than 10 units per litre of Anti-HBs.
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high risk group.
* In the opinion of the investigator, a subject who is not likely to complete the trial for what ever reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
To investigate genomic expression profiles after exposure to either intradermal avotermin (Juvista) or placebo | Days 3 and 5
To investigate the genomic expression profiles of reduced scarring in healthy male volunteers | Days 3 and 5 and month 6

SECONDARY OUTCOMES:
To collect further safety and toleration data for intradermal RN1001 | Day 15 and month 6
To assess systemic exposure following intradermal RN1001 before and after minor skin incisions | Day 15 and month 6
To confirm accelerated healing associated with intradermal RN1001 | Days 3 and 5
To investigate how to power a genomic analysis study optimally for the detection of gene expression profiles associated with accelerated healing, drug delivery and improved scarring. | Days 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Davies, Principal Investigator — Renovo; Jonathan Duncan, Principal Investigator — Renovo
Locations (1):
- Renovo Ltd, Manchester, United Kingdom